CLINICAL TRIAL: NCT04269252
Title: A Randomized Controlled Test of the Effects of CHI-907 on Experiences of Test Anxiety Among College Students
Brief Title: CHI-907 CBD Extract and Experiences of Test Anxiety
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment challenges due to COVID
Sponsor: Canopy Growth Corporation (Industry)
Collaborators: James Madison University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: USA710-4003
Record Dates: First submitted 2020-02-07; First posted 2020-02-13 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Anxiety
Keywords: Anxiety; Test Anxiety; CBD
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CHI-804 at 6 mL (Placebo Comparator): Standard 6 mL dose of placebo oil.
  Interventions: Other: CHI-804
- CHI-907 at 1.5 mL (Active Comparator): Subjects are assigned to receive one dose of CHI-907.
  Interventions: Other: CHI-907
- CHI-907 at 3 mL (Active Comparator): Subjects are assigned to receive one dose of CHI-907.
  Interventions: Other: CHI-907
- CHI-907 at 6 mL (Active Comparator): Subjects are assigned to receive one dose of CHI-907.
  Interventions: Other: CHI-907

INTERVENTIONS:
Other: CHI-907 — CHI-907 is a high CBD extract.
  Arms: CHI-907 at 1.5 mL; CHI-907 at 3 mL; CHI-907 at 6 mL
Other: CHI-804 — CHI-804 is the placebo formulation.
  Arms: CHI-804 at 6 mL

SUMMARY:
This is a randomized, placebo-controlled study examining the effects of CHI-907 on test anxiety specifically, and state anxiety more broadly.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult between 18 and 55-years-old (inclusive).
2. Willing and able to provide informed consent and attend a 2.5 hour, in-person session.
3. Self-reports completing a college-level introductory level statistics class with a grade of "C" or better.
4. Scores a 3.0 or higher on the Westside Test Anxiety Scale.
5. Female of childbearing potential must not be pregnant or currently breastfeeding.
6. If using medication, the student has maintained a stable regimen on existing medications for at least one month prior to participation in the study and throughout the study.
7. Agrees to abide by all study restrictions and comply with all study procedures.

Exclusion Criteria:

1. Known history of significant allergic condition, significant hypersensitivity to the IP, or allergic reaction to cannabis, cannabinoid medications, or excipients of the investigational product.
2. Exposed to any investigational drug or device < 30 days prior to screening or plans to take an investigational drug in the near future.
3. Used cannabis, synthetic cannabinoid or cannabinoid analogue, synthetic cannabinoid receptor agonist, or any CBD- or THC-containing product within 30 days of screening or during the study.
4. Current or past primary DSM-5 diagnosis other than an anxiety disorder that the Investigator determines would interfere in testing or interfere in evaluation of the study testing.
5. Total score of 8 or higher on the Alcohol Use Disorders Identification Test.
6. Total score of 12 or higher on the Drug Abuse Screening Test.
7. An acute or progressive disease that is likely to require changes in drug therapy during the study, or interfere with the objectives of the study, or the ability to adhere to protocol requirements.
8. Currently prescribed medications with likely THC- or CBD- interactions.
9. History of suicide attempt in the last year.
10. Endorses current suicidal intent during the baseline assessment.
11. Positive drug screen for THC, barbiturates, amphetamines, benzodiazepines, and/or opiates at baseline assessment.
12. Clinically significant condition or abnormal findings during screening or the baseline assessment that would, in the opinion of the Investigator, preclude study participation or interfere with the evaluation of the study testing.
13. Demonstrates behavior indicating unreliability or inability to comply with the requirements of the protocol.
14. Female student of childbearing potential, unless willing to ensure that they or their partner use effective contraception during the study and for three months thereafter.
15. Male student whose partner is of childbearing potential, unless willing to ensure that they or their partner use effective contraception during the study and for three months thereafter.
16. Any other significant disease or disorder which, in the opinion of the investigator, may either put the student at risk because of participation in the study, may influence the result of the study, or affect the student's ability to participate in the study.
17. History of diagnosis related to hepatic function and/or significantly impaired hepatic function (alanine aminotransferase [ALT] >5 ´ upper limit of normal [ULN] or total bilirubin [TBL] >2 ´ ULN) OR the ALT or aspartate aminotransferase (AST) >3 ´ ULN and TBL >2 ´ ULN (or international normalized ratio [INR] >1.5).
18. Plans for the student to travel outside their country of residence during the study.
19. Body mass index (BMI) of underweight (18 kg/m2 and below) or obese (30 kg/m2 and above) or waist:hip ratio that is considered high health risk (0.86 and higher for women, 1.0 and higher for men).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Optimal single-dose of CHI-907 to reduce test anxiety | The test session visit is 3.5 hours long.
  Subjects will report their level of test anxiety using the State Test Anxiety Visual Analog Scale (STAI-VAS) pre-test, mid-test, and post-test. The STAI-VAS is a measure from 0 (not anxious at all) to 100 (anxious).
Minimal single-dose of CHI-907 to reduce test anxiety | The test session visit is 3.5 hours long.
  Subjects will report their level of test anxiety using the State Test Anxiety Visual Analog Scale (STAI-VAS) pre-test, mid-test, and post-test. The STAI-VAS is a measure from 0 (not anxious at all) to 100 (anxious).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ware, MD, Study Director — Canopy Growth Corporation
Locations (1):
- James Madison University, Harrisonburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No